CLINICAL TRIAL: NCT06466382
Title: OV PRECISION: A Randomized Controlled Swiss Trial Examining the Benefit of a Tumor- and Patient-specific Cancer Therapy in Ovarian Cancer.
Brief Title: OV Precision: Study Examining the Benefit of a Tumor- and Patient-specific Cancer Therapy
Acronym: OVPrecision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss GO Trial Group (Network)
Collaborators: Tumor Profiler Center Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Swiss-GO-08/ OV Precision
Record Dates: First submitted 2024-05-21; First posted 2024-06-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Neoplasm Epithelial; Fallopian Tube Neoplasms; Ovarian Endometrioid Carcinoma; High-grade Serous Ovarian Carcinoma (HGSOC)
Keywords: Primary ovarian cancer (OC); Treatment naiive; Multi-modal tumor profiling; Treatment recommendation process; Multi-disciplinary tumor board; Patient benefit; Quality of Life (QoL); Patient-personalized therapy
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Physicians and patients randomized to the SOC arm will not receive the treatment recommendation of the mTB and thus will undergo the standard treatment consisting of 2 cycles of chemotherapy with carboplatin AUC5 3-weekly and paclitaxel 175 mg/m2 3-weekly or carboplatin AUC2 weekly and Paclitaxel 60-80mg/m2 weekly.
  Either q3w regime or q1w regime.
  Interventions: Drug: Carboplatin / Paclitaxel Chemotherapy
- Interventional Arm (Experimental): The intervention studied is a treatment recommendation by a specialized molecular tumorboard. This recommendation is based on an MSR which is created by TP, i.e., molecular analysis of clinical specimens, obtained from the individual participant. TP, a technology platform of several precision-cancer profiling domains, combines and rates the most efficient drugs/ experimental treatments for an individual ovarian cancer patient independent of standard of care. The usability in clinical practice of this recommendation will be tested. It should support the clinical decision of the treating oncologists and patients to choose the best possible therapy for the individual patient.
  Interventions: Other: Treatment recommendation by molecular tumorboard (mTB) based on tumor profiling

INTERVENTIONS:
Other: Treatment recommendation by molecular tumorboard (mTB) based on tumor profiling — The intervention studied is a treatment recommendation by a specialized molecular tumorboard (mTB). This recommendation is based on an MSR which is created by TP, i.e., molecular analysis of clinical specimens, obtained from the individual participant. TP, a technology platform of several precision-cancer profiling domains, combines and rates the most efficient drugs/ experimental treatments for an individual ovarian cancer patient independent of standard of care. The usability in clinical practice of this recommendation will be tested. It should support the clinical decision of the treating oncologists and patients to choose the best possible therapy for the individual patient.
  Arms: Interventional Arm
Drug: Carboplatin / Paclitaxel Chemotherapy — 2 cycles of chemotherapy with carboplatin AUC5 3-weekly and paclitaxel 175 mg/m2 3-weekly or carboplatin AUC2 weekly and Paclitaxel 60-80mg/m2 weekly
  Other Names: Standard of care chemotherapy regime
  Arms: Control Arm

SUMMARY:
The long-term goal of this research project is to demonstrate whether HRD negative (HPDneg) patients benefit when additional multi-modal biological tumor information is incorporated into the molecular tumor board (mTB) treatment recommendation process.

DETAILED DESCRIPTION:
Homologous recombination proficient (HRP) or HRD negative (HRDneg) Ovarian Cancer (OC) patients have a poor outcome equivalent to platinum-resistant patients (PFS 11.5 month). Given standard of care chemotherapy is not ideal for 50% of EOC and this patient population urgently needs alternative treatment options tailored to their individual tumor profile. Treatment options for the heterogeneous HRDneg patient group are scarce and mainly focus on symptom control and palliation, delaying time to symptomatic progression, and improving QoL.

Therefore, trials at initial diagnosis, when the patient can still be cured and is treatment naïve, are urgently needed.

The intervention studied is a personalized treatment recommendation by a specialized molecular tumorboard. This recommendation is based on a molecular summary report (MSR), which is created by multi-modal Tumor Profiling (TP), i.e., molecular analysis of clinical specimens, obtained from the individual participant.

TP, a technology platform of several precision-cancer profiling domains established by the TPC (= Tumor Profiler Center, Switzerland). It combines and rates the most efficient drugs/ experimental treatments for an individual ovarian cancer patient independent of standard of care (SOC).

The usability in clinical practice of this recommendation will be tested. It should support the clinical decision of the treating oncologists and patients to choose the best possible therapy for the individual patient. Treatment recommendations on the most appropriate molecular-based treatment for the individual patient are formulated based on the expertise and experience of the mTB board members. Additionally, a MSR from a validated TP technology platform can serve as further guidance in the tumorboard. However, the final decision on initial treatment remains at the discretion of the treating physician and the patient.

OV Precision is a multicenter randomized (1:1) controlled trial comparing a personalized treatment recommendation at the discretion of the treating physician in agreement with the patient versus SOC without receiving a mTB recommendation.

The study will be divided into two phases: an initial diagnostic phase, in which presumed eligible patients will be recruited into the study, HRD status will be determined, and tumor profiling will be performed in HRDneg patients with a confirmed diagnosis. Eligible patients will be randomized and treated according to their group allocation in the second phase (treatment phase).

The study duration is planned for 3 years including analysis: Two years of recruitment (starting from 09/2024), final analysis of the focal endpoints and end of the study 10 weeks after inclusion of the last patient (12/2026). Study analysis and publication should be completed approximately one year later (12/2027).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed EOC (adenocarcinoma of the ovary, peritoneum, and fallopian tube) and carcinosarcoma patients with a suspected FIGO Stage III and IV
* No immediate need of systemic or surgical treatment at time of and until 2 weeks after diagnosis
* Envisaged surgical candidate for interval debulking after 2 cycles of treatment
* Willing and able to attend the visits, to understand the purpose of the trial and all trial-related procedures
* ECOG 0-2
* Written informed consent according to national legal and regulatory requirements prior to any project specific procedures

Exclusion Criteria:

* Elevated liver enzymes (double of normal range: ASAT > 68 U/l; ALAT > 82 U/l; GGT > 80 U/l)
* Elevated creatinine (double of normal range: >120 mmol/l))
* ECOG ≥3
* Pregnant or lactating women
* Any other malignancy within the last 5 years which has an impact on the prognosis of the patient
* Inability to swallow tablets
* Concurrent participation in another clinical trial on the same indication
* Any other serious underlying medical, psychiatric, psychological, familial, or geographical condition, which in the judgment of the sponsor-project leader may interfere with the project or affect patient compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Focal Outcome Measure (FOM) 1 of pilot study: Proportion of patients for whom the molecular Tumor Board (mTB) considers a different treatment option | 2-3 weeks
  * Number (proportion) of cases in which the Tumor Profiling (TP) was able to generate a conclusive Molecular Summary Report (MSR)
  * Number (proportion) of cases in which the mTB considers the MSR as useful support for making a treatment recommendation on a scale from zero (not useful at all) to five (very useful)
FOM 2 of pilot study: Investigation whether the treating oncologist feels better supported by the mTB recommendation considers the additional biological tumor information than by the standard of care where such information is not considered. | 2-3 weeks
  * Number (proportion) of cases in which the treating physician considers the mTB recommendation as useful for making a final treatment decision on a scale from zero (not useful at all) to five (very useful).
  * Definition of molecular results from TP that cannot be used for clinical decision making.
  * Definition of an algorithm for the decision process from MSR to treatment recommendation.
FOM 3 of pilot study: Investigation of different treatment decisions by the patient and the treating oncologist. | 4 weeks
  * Number of therapy adaptations in the exploratory arm based on the MSR.
  * Number (proportion) of cases with therapy adaptions with minor / major/ no change from SOC.
  * Number (proportion) of treatment recommendations by mTB which were followed by the doctor and patient in the window of opportunity.
  * Number (proportion) of treatment recommendations by mTB which were continued by the doctor and patient after the trial and after finishing SOC.
  * Number (proportion) of treatment recommendations by mTB which were not followed by the doctor and patient in the window of opportunity due to restrictions.
  * Differences in hypothetical treatment costs between SOC and exploratory arm.
FOM 4 of pilot study: Preliminary estimate of the actual patient benefit of the intervention in terms of a number of patient-relevant outcomes. | 10 weeks
  The difference in proportions of responders between the standard of care and experimental arm after interval debulking surgery or biopsy at second specimen collection time point (week 10). A patient is classified as a responder if at least one of the two conditions is met: The Chemotherapy Response Score (CRS) is larger than or equal to 2 or the CA125 KELIM score is larger than or equal to 1.
  Note A : The three-tired CRS ranges from 1 (no or minimal tumor response) to 3 (total or near-total tumor response) .
  Note B: The tumormarker CA125 level decline (= CA125 KELIM ) over at least 3 timepoints can give an indication of therapy response. A favourable KELIM score ≥ 1.0, Unfavorable KELIM score < 1.
  * Symptoms measured by MOST- S26 questionnaire from V1 (baseline at diagnosis) until V9 (EOT), in both arms.
  * Quality of Life (QoL): Questionnaires EORTC QLQ-C30, EORTC QLQ-OV28 from V1 (baseline at diagnosis) until V9 (EOT), in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Viola Heinzelmann-Schwarz, Prof., Principal Investigator — University Hospital Basel, Head Women's Hospital
Locations (7):
- Switzerland (7):
  - Kantonsspital Baden AG, Baden, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - HOCH Health Ostschweiz Kantonsspital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Thurgau AG Frauenfeld / Münsterlingen, Frauenfeld, Thurgau
  - Inselspital Bern (University Hospital for Medical Oncology), Bern
  - HFR-Fribourg- Hopital Cantonal, Fribourg
  - University Hospital Zurich, Zurich